CLINICAL TRIAL: NCT00677690
Title: Combination of Pulmonary Rehabilitation and Neuromuscular Electrical Stimulation and in COPD Patients: a Randomized Clinical Trial of Efficacy
Brief Title: Neuromuscular Electrical Stimulation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Ercole Zanotti, MD, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2008
Record Dates: First submitted 2008-05-08; First posted 2008-05-14 (Estimated); Results first posted 2009-04-20 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NM+PR (Active Comparator): Patients undergone to combination of neuromuscular stimulation and pulmonary rehabilitation (NM+PR)
  Interventions: Other: neuromuscular electrical stimulation (NMES)
- SS+PR (Placebo Comparator): Patients undergone to pulmonary rehabilitation
  Interventions: Other: Sham electrical stimulation

INTERVENTIONS:
Other: neuromuscular electrical stimulation (NMES) — NMES was applied by means of a commercially available four channel electrostimulator which generated a symmetrical biphasic pulsed current. Each session lasted 30 minutes and was performed 5 days/week for 5 weeks.
  Other Names: pulmonary rehabilitation
  Arms: NM+PR
Other: Sham electrical stimulation — Sham stimulation was performed with the same modality and time, but the stimulus was set up at 5 Hz.
  Other Names: pulmonary rehabilitation
  Arms: SS+PR

SUMMARY:
The purpose of this study is to elucidate whether combination of usual pulmonary rehabilitation and neuromuscular electrical stimulation of quadriceps may improve exercise capacity in patients affected by chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation (NMES) has been extensively used as technique to improve muscle function in different areas of rehabilitation, however it seems to be more appropriate in critical care situation, while its use in more able patients is of uncertain benefit. In other words, NMES seems to be particularly effective in severely deconditioned and bed ridden patients. We therefore carried out a randomised trial to compare the efficacy of combination of NMES and PR (NM+PR) with combination of sham stimulation and PR (SS+PR) in a large population of moderately impaired COPD patients. Primary outcome was evaluation of effect of NMES on quadriceps strength and on exercise capacity. Secondary outcome was evaluation of effect of NMES on symptoms (dyspnoea) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Must be able to walk

Exclusion Criteria:

* Previous or current diagnosis of chronic respiratory failure
* A history of diseases other than COPD, in particular neurological disease
* Need for treatment with systemic steroids during the rehabilitation period

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ercole zanotti, MD, Principal Investigator — Fondazione Maugeri
Locations (1):
- Fondazione Salvatore Maugeri, Montescano, Pavia, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2007-2008 - Rehabilitative Pulmonary ward
Pre-assignment Details: 167 COPD patients were admitted.52 out of 167 did not meet the inclusion criteria.19 out of the remaining 115 patients refused to participate.13 out of 96 subjects subsequently dropped out due to acute exacerbation.Our definitive sample was therefore of 83 subjects
Groups:
- Neuromuscular Stimulation and Pulmonary Rehabilitation: Patients undergone to combination of neuromuscular stimulation and pulmonary rehabilitation
- Pulmonary Rehabilitation: Patients undergone to pulmonary rehabilitation
Period: Overall Study
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Started | 42 | 41
Completed | 42 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 31 | 32 | 63
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.6) | 62.8 (5.4) | 62.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 31 | 29 | 60
Region of Enrollment [Number; unit: participants]
  Italy | 42 | 41 | 83

OUTCOME MEASURES:

1. Secondary Outcome: Dyspnoea
Description: The modified Medical Research Council (MMRC) scale was used for rating dyspnoea. MMRC is a five-point scale based on degrees of various physical activities that precipitate breathlessness. Scores on the MMRC dyspnoea scale can range from 0 (normal) to 4.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Number analyzed (Participants) | 42 | 41
units on a scale | 2.4 (0.4) | 2.6 (0.2)
Statistical Analysis 1: Comparison: Neuromuscular Stimulation and Pulmonary Rehabilitation vs Pulmonary Rehabilitation; All data were expressed as the mean ± SD. The level of significance for all tests was set at p < 0.05. Inter- and intra-group comparisons were performed using both paired and unpaired t tests for continuous variables and Chi squared for categorical variables; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

2. Primary Outcome: Exercise Capacity
Description: 6 minute walk test(6MWT)
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Number analyzed (Participants) | 42 | 41
meters | 465.5 (101.7) | 462.7 (96.9)
Statistical Analysis 1: Comparison: Neuromuscular Stimulation and Pulmonary Rehabilitation vs Pulmonary Rehabilitation; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

3. Secondary Outcome: Quality of Life
Description: St. George's respiratory questionnaire is a standardized self-administered airways disease-specific questionnaire divided into three subscales: symptoms (eight items), activity (16 items), and impacts (26 items). For each subscale and for the overall questionnaire, scores range from zero (no impairment) to 100 (maximum impairment).
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Number analyzed (Participants) | 42 | 41
units on a scale | 41.7 (14.8) | 42.05 (15.7)
Statistical Analysis 1: Comparison: Neuromuscular Stimulation and Pulmonary Rehabilitation vs Pulmonary Rehabilitation; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

4. Primary Outcome: Quadriceps Strength
Description: Quadriceps strength was assessed by means of Sit to Stand Test (STST). The subjects held their arms stationary by putting their hands on their hips. The subjects were asked to complete the sitting and standing positions without using the arms for support while rising and sitting. Once instructed, subjects stand upright and without delay sit down again, repeating the procedure as many times as possible in a 1 min period. The number of completed repetitions was recorded. The subjects were permitted to use rest periods to complete 1 min.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Number analyzed (Participants) | 42 | 41
repetitions | 13.5 (0.83) | 13.6 (0.99)
Statistical Analysis 1: Comparison: Neuromuscular Stimulation and Pulmonary Rehabilitation vs Pulmonary Rehabilitation; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

5. Secondary Outcome: Respiratory Function
Description: forced expiratory volume in 1 second (FEV1)
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Number analyzed (Participants) | 42 | 41
percentage of predicted value | 50.1 (6.4) | 49.6 (8.2)
Statistical Analysis 1: Comparison: Neuromuscular Stimulation and Pulmonary Rehabilitation vs Pulmonary Rehabilitation; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Neuromuscular Stimulation and Pulmonary Rehabilitation | Pulmonary Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No